CLINICAL TRIAL: NCT03487744
Title: Comparison of the Incidence of Diarrhea Using High and Low Osmolality Enteral Tube Feeding in Critically Ill Surgical Patients
Brief Title: Incidence of Diarrhea Using High and Low Osmolality Enteral Tube Feeding in Critically Ill Surgical Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Amanda Zomp, Clinical Pharmacist, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB_00108798
Record Dates: First submitted 2018-03-20; First posted 2018-04-04 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Tube Feeding
Keywords: Tube Feeding; Diarrhea; Enteral Nutrition; Critically Ill; Surgical; Cardiovascular
MeSH Terms: conditions — Diarrhea; Critical Illness | interventions — Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Promote without fiber (Active Comparator): Lower osmolality enteral tube feed formulation
  Interventions: Other: Promote without fiber
- Osmolite 1.5 (Active Comparator): Higher osmolality enteral tube feed formulation
  Interventions: Other: Osmolite 1.5

INTERVENTIONS:
Other: Osmolite 1.5 — Continuous enteral tube feeding according to a standardized calculation via nasojejunal tube.
  Arms: Osmolite 1.5
Other: Promote without fiber — Continuous enteral tube feeding according to a standardized calculation via nasojejunal tube.
  Arms: Promote without fiber

SUMMARY:
The purpose and primary objective of this study is to determine if there is an association between enteral tube feed (TF) osmolality and diarrhea in critically ill patients. The investigators hypothesize that the administration of a TF formulation with high osmolality will cause more diarrhea than a TF formulation with a lower osmolality.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* admitted to SICU or CVICU requiring TF for enteral nutrition
* anticipated ICU stay and TF requirement >72 hours

Exclusion Criteria:

* Contraindication to receiving one of the study TF formulations
* Inability to tolerate at least 75% of estimated requirement by day 3 of enteral TF administration
* Clostridium difficile infection or other cause of infectious diarrhea prior to study enrollment
* Presence of an ileostomy or colostomy
* History of inflammatory bowel disease, bowel resection, short gut syndrome, or chronic diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of diarrhea at 72 hours | 72 hour

SECONDARY OUTCOMES:
Incidence of diarrhea at 14 days | 14 days
Mean frequency of diarrhea days | 14 days
Total number of diarrhea days | 14 days
Mean diarrhea scores | 14 days
  Hart and Dobb Diarrhea Scale (a tool based on consistency and size of each stool, with a sum of all stools in one day equaling the score for each day and a score of 12 or more indicates diarrhea)
Time at 75% or more of goal tube feeding rate | 14 days
Incidence of hypokalemia | 14 days
Incidence of perineal dermatitis | 14 days
Number of Clostridium difficile assays sent | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Health, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No